CLINICAL TRIAL: NCT03579680
Title: De-implementation of Low Value Castration for Men With Prostate Cancer
Acronym: DeADT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ted Skolarus, Adjunct Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00133932-1; 1R37CA222885-01 (NIH)
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Cancer of Prostate
Keywords: Prostatic Neoplasms; De-implementation; androgen deprivation therapy; Provider Preferences
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADT ORDER CHECK ATTESTATION (OR) (Experimental): Experimental: ADT ORDER CHECK ATTESTATION (OR) Order restrictions (Or) operate as an organizational constraint, widely perceived as a forcing function giving providers little leeway to exercise judgment but have a strong evidence-base for changing provider behavior. Study staff will place a "health factor" structured data element in the EMR of patients whose clinic visits study staff have confirmed to be targets for ADT de-implementation. This health factor combined with a low PSA level will trigger the ADT Order Check Attestation Intervention (Or) when the provider places an order for ADT.
  Interventions: Behavioral: ADT ORDER CHECK ATTESTATION (OR)
- PROVIDER SCRIPT (SC) (Experimental): Experimental: PROVIDER SCRIPT (SC) The provider script (Sc) is a communication aid to be used and documented as an accountable justification in the electronic medical record. This strategy also has a strong evidence-base for changing provider behavior. Study staff will enter a pre-populated CPRS EMR progress note 1 business day prior to a target clinic visit. The note includes talking points for the provider to help with a discussion. It can be edited and cosigned by the provider, giving a quick and simple way to document the discussion. The progress note template asks providers to indicate whether patient prefers to continue or discontinue low-value ADT. Appropriate documentation of the decision will be tracked for fidelity. We will also have a patient handout entitled: "Living well with prostate cancer: Is hormone therapy still right for you?" as a patient engagement and information resource.
  Interventions: Behavioral: PROVIDER SCRIPT (SC)

INTERVENTIONS:
Behavioral: ADT ORDER CHECK ATTESTATION (OR) — Order restrictions (Or) operate as an organizational constraint, widely perceived as a forcing function giving providers little leeway to exercise judgment but have a strong evidence-base for changing provider behavior.
  Arms: ADT ORDER CHECK ATTESTATION (OR)
Behavioral: PROVIDER SCRIPT (SC) — The provider script (Sc) is a communication aid to be used and documented as an accountable justification in the electronic medical record. This strategy also has a strong evidence-base for changing provider behavior.
  Arms: PROVIDER SCRIPT (SC)

SUMMARY:
This study will use a theory-based, mixed methods approach to identify, tailor and pilot two different de-implementation strategies that vary widely in delivery, impact, and expected results for reducing low value androgen deprivation therapy (ADT) use in preparation for a randomized comparative effectiveness trial comparing two tailored deimplementation strategies to reduce chemical castration as localized prostate cancer treatment and treatment for non-metastatic biochemical recurrence with low PSA levels.

DETAILED DESCRIPTION:
Prostate cancer is the leading cancer among Veterans. One in three Veterans with prostate cancer is chemically castrated at some point with long-acting injectable drugs (i.e., androgen deprivation therapy, or ADT). This impacts the well-being of thousands of Veterans annually. Although some patients benefit in terms of survival and symptom improvement, chemical castration with ADT is also commonly performed when there are little to no health benefits to patients raising questions of low value care. A growing awareness of castration harms (e.g., heart attack, osteoporosis, loss of sexual function) creates patient safety concerns. Despite this, ADT use in low value cases, such as for localized prostate cancer treatment, persists in the Veterans Health Administration (VHA) with five-fold variation across its facilities. Ineffective and harmful practices such as chemical castration of prostate cancer patients with ADT outside of the evidence base are ideal targets for de-implementation. De-implementation, or stopping low value practices, has the potential to improve patient outcomes and decrease healthcare costs. However, provider preferences regarding de-implementation are not well understood, and possible de-implementation interventions range from blunt formulary restriction policies to informed decision-making. Both intervention strategies need tailoring based on provider input for acceptability and feasibility in clinical practice, including piloting prior to trialing. As many medical practices lack evidence and cause harm, robust, behavioral theory-based methods for incorporating provider preferences into de-implementation strategy development will advance both implementation research and practice.

This study will use a theory-based, mixed methods approach to identify, tailor and pilot two different de-implementation strategies that vary widely in delivery, impact, and expected results for reducing low value ADT use, in preparation for a randomized comparative effectiveness trial.

This innovative mixed-methods research program has three aims, of which Aim 3 is represented in this registration.

Aim 1: To assess preferences and barriers for de-implementation of chemical castration in prostate cancer. Guided by the Theoretical Domains Framework (TDF), urologists and patients from facilities with the highest and lowest castration rates across VHA will be interviewed to identify key preferences and deimplementation barriers for reducing castration as prostate cancer treatment. This qualitative work will inform Aim 2 while gathering rich information for two proposed pilot intervention strategies.

Aim 2: To use a discrete choice experiment (DCE), a novel barrier prioritization approach, for deimplementation strategy tailoring. The investigators will conduct national surveys of US Government urologists to prioritize key barriers identified in Aim

1 for stopping incident castration as localized prostate cancer treatment using a discrete choice experiment design. These quantitative results will identify the most important barriers to be addressed through tailoring of two pilot deimplementation strategies in preparation for Aim 3 piloting.

Aim 3: To pilot two tailored de-implementation strategies to reduce castration as localized prostate cancer treatment and treatment for non-metastatic biochemical recurrence with low PSA levels. Building on findings from Aims 1 and 2, two de-implementation strategies will be piloted. One strategy will focus on formulary restriction/ order check attestation at the organizational level and the other on physician/ patient informed decision-making at different facilities. Pilot outcomes will include feasibility at the site level, feasibility at the clinic level, reach, and penetration in preparation for an effectiveness trial comparing these two widely varying de-implementation strategies. This innovative approach to de-implementation strategy development will transform how and why castration is performed for localized prostate cancer and nonmetastatic biochemical recurrence with low PSA levels through combining provider and patient preferences and strategy tailoring. This work will advance de-implementation science for low value care and foster participation in a subsequent de-implementation evaluation trial by addressing barriers, facilitators and concerns through pilot tailoring.

ELIGIBILITY:
Inclusion Criteria:

- Any provider at participating sites who prescribes ADT for prostate cancer patients

Exclusion Criteria:

- Providers opting out of study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2023-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ted Skolarus, MD, Principal Investigator — University of Michigan/Department of Veterans Affairs
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Members of the scientific community who would like a copy of the de-identified final data sets (i.e., data sets underlying any publication) from this study can request a copy by e-mailing Jennifer Burns at jennifer.burns@va.gov. They should state their reason for requesting the data and their plans for analyzing the data. Final data sets will be copied onto an encrypted CD. The CD will be sent to the requestor via FedEx.
Time Frame: Data will be available once pilot is complete and up to 6 years after the end of the fiscal year in which the project is terminated.
Access Criteria: Members of the scientific community who would like a copy of the de-identified final data sets (i.e., data sets underlying any publication) from this study can request a copy by e-mailing Jennifer Burns at jennifer.burns@va.gov. They should state their reason for requesting the data and their plans for analyzing the data. Final data sets will be copied onto an encrypted CD. The CD will be sent to the requestor via FedEx.

REFERENCES:
- [Derived] Skolarus TA, Hawley ST, Forman J, Sales AE, Sparks JB, Metreger T, Burns J, Caram MV, Radhakrishnan A, Dossett LA, Makarov DV, Leppert JT, Shelton JB, Stensland KD, Dunsmore J, Maclennan S, Saini S, Hollenbeck BK, Shahinian V, Wittmann DA, Deolankar V, Sriram S. Unpacking overuse of androgen deprivation therapy for prostate cancer to inform de-implementation strategies. Implement Sci Commun. 2024 Apr 9;5(1):37. doi: 10.1186/s43058-024-00576-x. PMID 38594740
- [Derived] Skolarus TA, Forman J, Sparks JB, Metreger T, Hawley ST, Caram MV, Dossett L, Paniagua-Cruz A, Makarov DV, Leppert JT, Shelton JB, Stensland KD, Hollenbeck BK, Shahinian V, Sales AE, Wittmann DA. Learning from the "tail end" of de-implementation: the case of chemical castration for localized prostate cancer. Implement Sci Commun. 2021 Oct 28;2(1):124. doi: 10.1186/s43058-021-00224-8. PMID 34711274
- [Derived] Skolarus TA, Hawley ST, Wittmann DA, Forman J, Metreger T, Sparks JB, Zhu K, Caram MEV, Hollenbeck BK, Makarov DV, Leppert JT, Shelton JB, Shahinian V, Srinivasaraghavan S, Sales AE. De-implementation of low value castration for men with prostate cancer: protocol for a theory-based, mixed methods approach to minimizing low value androgen deprivation therapy (DeADT). Implement Sci. 2018 Nov 29;13(1):144. doi: 10.1186/s13012-018-0833-7. PMID 30486836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Providers (physicians) had the option to opt out of the study.
Units Other Than Participants: Centers
Groups:
- ADT ORDER CHECK ATTESTATION (OR): Experimental:
  ADT ORDER CHECK ATTESTATION (OR): Order restrictions (Or) operate as an organizational constraint, widely perceived as a forcing function giving providers little leeway to exercise judgment but have a strong evidence-base for changing provider behavior.
  (In some publications, this is also referred to as Clinical Reminder Order Check (CROC).)
Period: Overall Study
Arm/Group | ADT ORDER CHECK ATTESTATION (OR) | PROVIDER SCRIPT (SC)
Started | 46; 3 Centers | 14; 1 Centers
Completed (One center was not able to fully operationalize the electronic health record (CPRS) intervention due to informatics, regulatory, and workforce delays.) | 46; 2 Centers (Of all physicians involved, none opted out, but one center couldn't fully implement the project.) | 14; 1 Centers
Not Completed | 0; 1 Centers | 0; 0 Centers

BASELINE CHARACTERISTICS:
Population: No demographic data was collected on physician participants, nor on the patients they treated. Neither of these two groups required consenting. Only site/center level approval was obtained.
Groups:
- Total: Total of all reporting groups
Arm/Group | ADT ORDER CHECK ATTESTATION (OR) | PROVIDER SCRIPT (SC) | Total
Number analyzed (Participants) | 46 | 14 | 60
Age, Customized [Count of Participants; unit: Participants] — No age data was gathered, but all clinicians were adults.
  Participants
    All clinicians were adults > age 18; | 46 | 14 | 60
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex, gender of the physicians was not collected or studied. All of the patients affected were male as the study was looking at de-implementation of androgen deprivation therapy (ADT) injections. But no patient level demographic data was gathered for this feasibility trial.
  The sites which were the unit of measure of interest, and at which the trial was conducted have no gender, race, ethnicity or biological age. Population: No gender/sex data was collected on the providers/clinicians
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46 | 14 | 60

OUTCOME MEASURES:

1. Primary Outcome: Feasibility - Site Level: Medical Center Director (MCD) Approval
Description: The percentage of pilot sites asked to participate that received MCD approval to implement the intervention (Order Check or Progress Note/Patient Handout)
Time Frame: Within 1 month
Measure: Count of Units; unit: sites
Units Other Than Participants: sites
Groups:
- ADT ORDER CHECK ATTESTATION (OR): ADT ORDER CHECK ATTESTATION (OR) Order restrictions (Or) operate as an organizational constraint, widely perceived as a forcing function giving providers little leeway to exercise judgment but have a strong evidence-base for changing provider behavior.
  (In some publications, this is also referred to as Clinical Reminder Order Check (CROC).)
Arm/Group | ADT ORDER CHECK ATTESTATION (OR) | PROVIDER SCRIPT (SC)
Number analyzed (Participants) | 46 | 14
Number analyzed (sites) | 3 | 1
sites | 3 | 1

2. Primary Outcome: Feasibility - Site Level: Fully Operationalized Intervention
Description: The percentage of approved pilot sites with fully operationalized intervention, i.e. intervention successfully programmed into site Electronic Health Records and ready to be implemented. Depending on randomization arm, this includes either health factor placement or script assignment prior to at least one patient visit.
Time Frame: Within 6 months of approval
Measure: Count of Units; unit: sites
Units Other Than Participants: sites
Arm/Group | ADT ORDER CHECK ATTESTATION (OR) | PROVIDER SCRIPT (SC)
Number analyzed (Participants) | 46 | 14
Number analyzed (sites) | 3 | 1
sites | 2 | 1

3. Primary Outcome: Feasibility - Clinic Level: Clinics With Intervention Implementation
Description: The percentage of clinics at approved pilot sites with at least 1 intervention implemented, i.e. at least 1 health factor assigned and/or at least 1 progress note assigned to a provider. Clinics may include Urology, Medical Oncology, and Radiation Oncology.
Time Frame: Within 6 months of intervention implementation
Population: While providers represented the "participants" for the purposes of participating or opting out, the relevant measure for this outcome is "sites".
Measure: Count of Units; unit: sites
Units Other Than Participants: sites
Arm/Group | ADT ORDER CHECK ATTESTATION (OR) | PROVIDER SCRIPT (SC)
Number analyzed (Participants) | 46 | 14
Number analyzed (sites) | 3 | 1
sites | 2 | 1

4. Secondary Outcome: Reach
Description: The percentage of providers prescribing ADT for prostate cancer sent an information sheet who did not opt out of the study.
Time Frame: Within 6 months of intervention
Population: Here participants are actually providers
Measure: Count of Participants; unit: Participants
Groups:
- ADT ORDER CHECK ATTESTATION (OR): Experimental: ADT ORDER CHECK ATTESTATION (OR): Order restrictions (Or) operate as an organizational constraint, widely perceived as a forcing function giving providers little leeway to exercise judgment but have a strong evidence-base for changing provider behavior.
  (In some publications, this is also referred to as Clinical Reminder Order Check (CROC).)
  (In some publications, this is also referred to as Clinical Reminder Order Check (CROC).)
Arm/Group | ADT ORDER CHECK ATTESTATION (OR) | PROVIDER SCRIPT (SC)
Number analyzed (Participants) | 46 | 14
Participants | 46 | 14

5. Secondary Outcome: Penetration - Provider Script (SC)
Description: Percentage of SC intervention clinic notes assigned to providers that were signed.
Time Frame: Within 6 months of intervention
Population: For this outcome measure, the number of providers at the site that adopted provider script is not considered. This outcome measure looks at the percentage of notes that were signed by a provider, but not the number of providers that signed notes.
Measure: Count of Units; unit: notes
Units Other Than Participants: notes
Arm/Group | PROVIDER SCRIPT (SC)
Number analyzed (Participants) | 14
Number analyzed (notes) | 8
notes | 5

6. Secondary Outcome: Penetration - OR
Description: Percentage of OR intervention order checks justified.
Time Frame: Within 6 months of intervention
Population: For this outcome measure the number of providers at the sites that used ADT order check attestation is not considered. This outcome measure is simply looking at the percent of order checks that were justified by the provider.
Measure: Count of Units; unit: orders checked
Units Other Than Participants: orders checked
Arm/Group | ADT ORDER CHECK ATTESTATION (OR)
Number analyzed (Participants) | 46
Number analyzed (orders checked) | 12
orders checked | 8

ADVERSE EVENTS:
Time Frame: Clinic participation was approximately six months long but no AE data was collected.
Description: No AE data was collected in any form - as this was just a feasibility study for implementation.
Groups:
- ADT ORDER CHECK ATTESTATION (OR): Experimental: ADT ORDER CHECK ATTESTATION (OR) Order restrictions (Or) operate as an organizational constraint, widely perceived as a forcing function giving providers little leeway to exercise judgment but have a strong evidence-base for changing provider behavior.
- PROVIDER SCRIPT (SC): Experimental: PROVIDER SCRIPT (SC) The provider script (Sc) is a communication aid to be used and documented as an accountable justification in the electronic medical record. This strategy also has a strong evidence-base for changing provider behavior.
Arm/Group | ADT ORDER CHECK ATTESTATION (OR) | PROVIDER SCRIPT (SC)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT03579680/Prot_SAP_000.pdf